CLINICAL TRIAL: NCT05327790
Title: A Dual-center, Double Blind, Randomized Placebo-controlled Pilot Trial of Concomitant Lyophilized Fecal Microbiota Transplantation (LFMT) and Biologic Therapy (Vedolizumab or Ustekinumab) for the Induction of Remission in Ulcerative Colitis (UC)
Brief Title: LFMT vs Placebo in New Biologic Start for Ulcerative Colitis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00117170
Record Dates: First submitted 2022-03-25; First posted 2022-04-14 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Ulcerative Colitis
Keywords: FMT; Microbiome
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: To maintain blinding, LFMT and placebo capsules will appear identical.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- LFMT capsules + vedolizumab (Experimental): The initial loading dose is 15 capsules, administered on day 0, in the clinic under direct observation, followed by 5 capsules daily starting on day 1 for 8 weeks at home. All subsequent doses will be dispensed to participants.
  Interventions: Drug: Lyophilized fecal microbiota (LFMT)
- Placebo capsules + vedolizumab (Placebo Comparator): The placebo capsules will appear identical to the LFMT capsules; however, the capsules will contain 2 ingredients: trehalose and neusilin, which are components in LFMT capsules.
  Interventions: Other: Placebo
- LFMT capsules + ustekinumab (Experimental): The initial loading dose is 15 capsules, administered on day 0, in the clinic under direct observation, followed by 5 capsules daily starting on day 1 for 8 weeks at home. All subsequent doses will be dispensed to participants.
  Interventions: Drug: Lyophilized fecal microbiota (LFMT)
- Placebo capsules + ustekinumab (Placebo Comparator): The placebo capsules will appear identical to the LFMT capsules; however, the capsules will contain 2 ingredients: trehalose and neusilin, which are components in LFMT capsules.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Lyophilized fecal microbiota (LFMT) — vedolizumab or ustekinumab + FMT vs placebo
  Arms: LFMT capsules + ustekinumab; LFMT capsules + vedolizumab
Other: Placebo — Placebo
  Arms: Placebo capsules + ustekinumab; Placebo capsules + vedolizumab

SUMMARY:
To compare the safety and efficacy of concomitant LFMT versus placebo in UC patients who are starting vedolizumab or ustekinumab.

DETAILED DESCRIPTION:
This is dual-center, randomized, double-blind, placebo-controlled pilot trial for UC patients with active disease who are being initiated on treatment with vedolizumab or ustekinumab.

The study will recruit 40 outpatients at 2 Canadian healthcare centres at the University of Alberta Hospital (University of Alberta), and the University of Manitoba.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older but less than 75 years of age
2. Able to provide informed consent
3. Established ulcerative colitis diagnosis determined by a physician through standard endoscopic and histologic criteria
4. Active UC defined as total Mayo score between 6-12 AND Mayo endoscopic sub-score >1 with disease that extends 15 cm or more from the anal verge
5. Selected by treating physician for initiation of biologic treatment with either vedolizumab or ustekinumab. Patients must be:

   * Biologic naive; OR
   * Have failed anti-TNF, anti-integrin, anti IL12/23 or oral small molecules
6. Use of effective contraception method for women of childbearing potential for at least 4 weeks prior to receiving study treatment and for the duration of the trial
7. Willing and able to comply with all required study procedures

Exclusion Criteria:

1. Severe UC requiring hospitalization
2. Indeterminate colitis
3. Evidence of or treatment for C difficile infection or other intestinal pathogen, including CMV, within 4 weeks prior to enrollment
4. Evidence of toxic megacolon or gastrointestinal perforation on imaging
5. Abdominal surgery within the past 60 days

   * Neutropenia with absolute neutrophil count <0.5 x 109/L
   * Peripheral white blood cell count > 35.0 x 109/L and fever (>38 degrees Celsius)
   * Planned or actively taking another investigational product
   * Uncontrolled medical conditions such as psychiatric disorders or substance abuse
   * Severe underlying disease such that the patient is not expected to survive for at least 30 days
6. Pregnant or lactating
7. Unwilling to discontinue non-dietary probiotic
8. Antibiotic use in the past 30 days or anticipated need for systemic antibiotic use during study
9. FMT within 3 months prior to enrollment
10. Use of the following medications:

    1. rectal/topical therapy within 2 weeks of screening
    2. cyclosporine, tacrolimus or thalidomide within 4 weeks of screening
    3. tofacitinib within 4 weeks of screening
    4. adalimumab or infliximab within 8 weeks of screening
    5. vedolizumab within 8 weeks of screening
    6. ustekinumab within 12 weeks of screening
    7. prednisone > 30 mg/d
11. Investigator deems enrolment in the study is not in the best interest of the patient

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-06-03 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with serious adverse events (SAEs) of interest up to week 8 in each group (ie vedolizumab with or without LFMT, ustekinumab with or without LFMT). | 24 weeks
  SAE of interest is defined as one of the following:
  * An infection attributable to FMT
  * Worsening UC, defined as requiring rescue therapy such as increase in steroid dose or change in biologic or colectomy
  * Hospitalization due to UC or an infection attributable to FMT
  * Mortality due to UC or an infection attributable to FMT
  SAE of interest is defined as one of the following:
  * An infection attributable to FMT
  * Worsening UC, defined as requiring rescue therapy such as increase in steroid dose or change in biologic or colectomy
  * Hospitalization due to UC or an infection attributable to FMT
  * Mortality due to UC or an infection attributable to FMT

SECONDARY OUTCOMES:
Proportion of participants in each group with adverse events during the study up to week 24, including nausea, vomiting, abdominal pain, worsening diarrhea, constipation or fevers | 24 weeks
Proportion of participants who achieve clinical remission, defined as total Mayo score ≤ 2 with no individual subscore > 1, at week 8 and 24 in each group. | 24 weeks
Proportion of participants who achieve clinical response | 24 weeks
  Defined as a reduction in the Mayo clinic score of ≥ 3 points and/ or ≥ 30% from baseline, with a decrease in the rectal bleeding subscore of ≥ 1 point or a subscore ≤ 1 at week 8 and 24 in each group
Proportion of participants who achieve symptom remission, defined as partial Mayo score < 2 with no individual subscore > 1, at week 8 and 24 in each group | 24 weeks
Proportion of participants who achieve symptom response, defined as reduction in partial Mayo score ≥ 2 points from baseline and ≥ 30% from baseline and decrease in rectal bleeding score of ≥ 1point from baseline, at week 8 and 24 in each group | 24 weeks
Proportion of participants who achieve endoscopic improvement, defined as Mayo endoscopic subscore ≤1, at week 8 and 24 in each group | 24 weeks
Changes in partial Mayo score over time up to week 24 relative to baseline in each group | 24 weeks
Changes in quality of life, assessed by short IBD Questionnaire (sIBDQ), and work productivity, assessed by Work Productivity and Activity Impairment Questionnaire (WPAIQ), at week 8 and 24 relative to baseline in each group | 24 weeks
Changes in inflammatory markers (serum c-reactive protein (CRP) and fecal calprotectin) over time up to week 24 in each group | 24 weeks

OTHER OUTCOMES:
Proportion of participants with Corticosteroid-free remission at week 8 and 24 | 24 weeks
Time to clinical remission, clinical response, symptom remission and symptom response in each group | 24 weeks
Changes in stool microbiome at week 8 and 24 relative to baseline in each group | 24 weeks
Changes in stool microbiome at time of remission relative to baseline in each group | 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No